## Table 1. Research Workflow

## PRELIMINARY PROCESS

Obtaining permissions for scales, Literature research, Preparation of training program, Receiving expert opinions, Obtaining the permissions of the ethics committee and institution,

## IMPLEMENTATION STAGE

(9,10,11. Class Student)

Sample creation: Taking the height and weight, body mass indexes of 1300 female students and reaching the sample group. Obtaining family and individual consent

